CLINICAL TRIAL: NCT01256593
Title: DRUG USE INVESTIGATION OF LYRICA(REGULATORY POST MARKETING COMMITMENT PLAN)
Brief Title: Safety And Efficacy Of Lyrica (Regulatory Post Marketing Commitment Plan)
Acronym: RAINBOW
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A0081261
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-08

CONDITIONS: Neuralgia
Keywords: Lyrica; Regulatory Post Marketing Commitment Plan; Safety; Neuropathic Pain; Post Marketing Surveillance
MeSH Terms: conditions — Neuralgia | interventions — Pregabalin; Capsules

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregabalin (Lyrica) capsule: Patients administered "Pregabalin capsule".
  Interventions: Drug: Pregabalin (Lyrica) capsule

INTERVENTIONS:
Drug: Pregabalin (Lyrica) capsule — Lyrica® Capsules depending on the investigator prescription. Frequency and duration are according to Package Insert as follows. "The usual adult dosage for oral use begins at 150 mg/day of pregabalin in twice daily, and should be gradually increased to 300 mg/day over 1 week or more and should be orally administered twice daily. Dosage should be adjusted, depending on age or symptoms. However, the daily maximum dose should not be beyond 600 mg, and should be orally administered twice daily".
  Other Names: Lyrica® Capsules 25 mg, Lyrica® Capsules 75 mg, Lyrica® Capsules 150 mg

SUMMARY:
The objective of this Investigation is to evaluate the safety and efficacy of Lyrica in medical practice. Also, occurrence of unknown and known adverse drug reactions (ADRs) in subjects treated with Lyrica will be monitored during the survey period, and whether an additional treatment outcome investigation and/or a post-marketing clinical study is required in the future will be determined.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes the first Lyrica® should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

* Patients need to be administered Lyrica® in order to be enrolled in the surveillance.

Exclusion Criteria:

* Patients not administered Lyrica®.

Min Age: 0 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involving A0081261 prescribes the Lyrica capsule.
Sampling Method: Probability Sample
Enrollment: 3827 (Actual)
Dates: Start 2011-02-05 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081261&StudyName=Safety%20And%20Efficacy%20Of%20Lyrica%20%28Regulatory%20Post%20Marketing%20Commitment%20Plan%29

RESULTS

PARTICIPANT FLOW:
Groups:
- LYRICA Capsules (Pregabalin): Participants who received LYRICA Capsules as indicated in the approved local product document were observed for a period of 13 weeks at maximum. The dosage can be adjusted as per physician's discretion.
Period: Overall Study
Arm/Group | LYRICA Capsules (Pregabalin)
Started | 3827
Completed | 3613 (Number of participants whose survey form were collected and included in analyses is shown.)
Not Completed | 214
Not completed — Protocol Violation | 26
Not completed — No Drug Administration Information | 2
Not completed — No Visit After Treatment | 186

BASELINE CHARACTERISTICS:
Population: Among 3827 participants whose survey form was collected, a total of 214 participants were excluded from the baseline analysis population due to following reasons: protocol violation (26 participants), no drug administration information (2 participants), and no visit after treatment (186 participants).
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 3613
Age, Customized [Number; unit: Participants]
  <15 years | 3
  ≥15 and <65 years | 1330
  ≥65 years | 2280
Sex/Gender, Customized [Number; unit: Participants]
  Male | 1684
  Female | 1929
Race/Ethnicity, Customized [Number; unit: Participants]
  Race and Ethnicity Not Collected | 3613

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Drug Reaction
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to LYRICA Capsules in a participant who received LYRICA Capsules. Relatedness to LYRICA Capsules was assessed by the physician.
Time Frame: 13 weeks at maximum
Population: The analysis population for this outcome measure was the baseline analysis population, which comprised of participants who satisfied the criteria of safety analysis population and had received LYRICA Capsules at least once.
Measure: Number; unit: Percentage of Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 3613
Percentage of Participants | 15.03

2. Secondary Outcome: Percentage of Participants With Serious Adverse Drug Reaction
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to LYRICA Capsules in a participant who received LYRICA Capsules. A serious ADR was an ADR resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Relatedness to LYRICA Capsules was assessed by the physician.
Time Frame: 13 weeks at maximum
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 3613
Percentage of Participants | 0.61

3. Secondary Outcome: The Percentage of Participants With Adverse Drug Reaction Unexpected From Japanese Package Insert
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to LYRICA Capsules in a participant who received LYRICA Capsules. Expectedness of the adverse event was determined according to the Japanese package insert. Relatedness to LYRICA Capsules was assessed by the physician.
Time Frame: 13 weeks at maximum
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 3613
Percentage of Participants | 0.42

4. Secondary Outcome: Number of Participants With Adverse Drug Reactions Related to Peripheral Edema or Other Edema-related Events
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to LYRICA Capsules in a participant who received LYRICA Capsules. Relatedness to LYRICA Capsules was assessed by the physician. Occurrence of ADRs related to peripheral edema or other edema-related events was evaluated.
Time Frame: 13 weeks at maximum
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 3613
Participants | 53

5. Secondary Outcome: Number of Participants With Adverse Drug Reactions Related to Dizziness, Somnolence, Loss of Consciousness, Syncope, and Potential for Accidental Injury
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to LYRICA Capsules in a participant who received LYRICA Capsules. Relatedness to LYRICA Capsules was assessed by the physician. Occurrence of ADRs related to dizziness, somnolence, loss of consciousness, syncope, and potential for accidental injury was evaluated.
Time Frame: 13 weeks at maximum
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 3613
Participants | 351

6. Secondary Outcome: Number of Participants With Adverse Drug Reactions Related to Vision-related Events
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to LYRICA Capsules in a participant who received LYRICA Capsules. Relatedness to LYRICA Capsules was assessed by the physician. Occurrence of ADRs related to vision-related events was evaluated.
Time Frame: 13 weeks at maximum
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 3613
Participants | 16

7. Secondary Outcome: Clinical Effectiveness Rate
Description: Clinical effectiveness of LYRICA Capsules was determined by the physician based on the following categories: (1) effective, (2) ineffective, or (3) impossible to judge at Week 13 of the treatment. Clinical effectiveness rate, which was defined as the percentage of participants who achieved clinical effectiveness over the total number of the analysis population, was presented along with the corresponding 2-sided 95% CI. For the participants who completed or discontinued the treatment before Week 13, the data at the time of the completion or discontinuation was used for the analysis.
Time Frame: At Week 13
Population: The analysis population for this outcome measure comprised of participants for whom the evaluation outcome of clinical effectiveness was available and who satisfied the inclusion criteria among the baseline analysis population. Of these, participants evaluated as "impossible to judge" were excluded from the analysis population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 3567
Percentage of Participants | 84.1 [82.8 to 85.3]

8. Secondary Outcome: Change From Baseline in Participant-rated Pain Score at Week 13
Description: The pain experienced at Week 13 during the past 24 hours was rated by participants at the time of getting up in the morning on an 11-grade scale, ranging from 0 (no pain) to 10 (the most severe pain possible). Mean change from baseline in participant-rated pain score at Week 13 was presented along with standard deviation. For the participants who completed or discontinued the treatment before Week 13, the data at the time of the completion or discontinuation was used for the analysis.
Time Frame: Baseline and at Week 13
Population: The analysis population for this outcome measure comprised of participants for whom the evaluation outcome of participant-rated pain score was available and who satisfied the inclusion criteria among the baseline analysis population.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 1843
Units on a scale | -3.4 (2.61)

9. Secondary Outcome: Change From Baseline in Participant-rated Sleep Interference Score at Week 13
Description: The sleep interference (inability to sleep because of pain) experienced at Week 13 during the past 24 hours was rated by participants at the time of getting up in the morning on an 11-grade scale, ranging from 0 (no disturbance) to 10 (totally unable to sleep because of pain). Mean change from baseline in participant-rated sleep interference score at Week 13 was presented along with standard deviation. For the participants who completed or discontinued the treatment before Week 13, the data at the time of the completion or discontinuation was used for the analysis.
Time Frame: Baseline and at Week 13
Population: The analysis population for this outcome measure comprised of participants for whom the evaluation outcome of participant-rated sleep interference score was available and who satisfied the inclusion criteria among the baseline analysis population.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 1550
Units on a scale | -2.4 (2.90)

10. Secondary Outcome: Patient's Impression (PGIC) at Week 13
Description: The patient's impression (patient global impression of change [PGIC]) at Week 13, as compared to the baseline condition (including the first day of treatment), was rated by participants on a 7-grade scale. For the participants who completed or discontinued the treatment before Week 13, the data at the time of the completion or discontinuation was used for the analysis.
Time Frame: At Week 13
Population: The analysis population for this outcome measure comprised of participants for whom the evaluation outcome of PGIC was available and who satisfied the inclusion criteria among the baseline analysis population.
Measure: Number; unit: Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 3567
Participants
  Markedly improved | 583
  Improved | 1039
  Slightly improved | 708
  Unchanged | 454
  Slightly worsened | 12
  Worsened | 11
  Markedly worsened | 1
  Not assessed | 759

11. Secondary Outcome: Physician's Impression (CGIC) at Week 13
Description: The physician's impression (clinical global impression of change [CGIC]) at Week 13, as compared to the baseline condition (including the first day of treatment), was rated by the physician on a 7-grade scale. For the participants who completed or discontinued the treatment before Week 13, the data at the time of the completion or discontinuation was used for the analysis.
Time Frame: At Week 13
Population: The analysis population for this outcome measure comprised of participants for whom the evaluation outcome of CGIC was available and who satisfied the inclusion criteria among the baseline analysis population.
Measure: Number; unit: Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 3567
Participants
  Markedly improved | 626
  Improved | 1149
  Slightly improved | 773
  Unchanged | 471
  Slightly worsened | 9
  Worsened | 6
  Markedly worsened | 1
  Not assessed | 532

ADVERSE EVENTS:
Time Frame: 13 weeks at maximum
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both serious and non-serious events during the study.
Arm/Group | LYRICA Capsules (Pregabalin)
All-Cause Mortality (participants affected / at risk) | 17/3613
Serious Adverse Events (participants affected / at risk) | 77/3613
Other Adverse Events (participants affected / at risk) | 636/3613
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LYRICA Capsules (Pregabalin) (N=3613)
Gangrene (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 1
Herpes zoster oticus (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Lymphangitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 6
Septic shock (Infections and infestations) | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Decreased immune responsiveness (Immune system disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hallucination (Psychiatric disorders) | 1
Hallucination, auditory (Psychiatric disorders) | 1
Somatic symptom disorder (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Altered state of consciousness (Nervous system disorders) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 11
Haemorrhagic cerebral infarction (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Paraparesis (Nervous system disorders) | 1
Radiculopathy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 3
Conjunctival haemorrhage (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 2
Arrhythmia (Cardiac disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Anorectal disorder (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Bladder disorder (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Condition aggravated (General disorders) | 1
Death (General disorders) | 1
Disease progression (General disorders) | 7
Drug interaction (General disorders) | 1
Generalised oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Oedema (General disorders) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 4
Femur fracture (Injury, poisoning and procedural complications) | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 3
Thermal burn (Injury, poisoning and procedural complications) | 1
Device breakage (Product Issues) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LYRICA Capsules (Pregabalin) (N=3613)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Sinus bradycardia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 27
Abnormal sensation in eye (Eye disorders) | 1
Accommodation disorder (Eye disorders) | 1
Dacryostenosis acquired (Eye disorders) | 1
Diabetic retinopathy (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Photophobia (Eye disorders) | 1
Photopsia (Eye disorders) | 1
Vision blurred (Eye disorders) | 10
Visual acuity reduced (Eye disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 3
Cheilitis (Gastrointestinal disorders) | 1
Chronic gastritis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 33
Diarrhoea (Gastrointestinal disorders) | 7
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 3
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Intestinal obstruction (Gastrointestinal disorders) | 1
Lip swelling (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 27
Oesophagitis (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 6
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Chills (General disorders) | 1
Discomfort (General disorders) | 1
Face oedema (General disorders) | 8
Feeling abnormal (General disorders) | 11
Feeling hot (General disorders) | 1
Gait disturbance (General disorders) | 2
Loss of control of legs (General disorders) | 1
Malaise (General disorders) | 4
Oedema (General disorders) | 26
Oedema due to cardiac disease (General disorders) | 2
Oedema peripheral (General disorders) | 37
Pain (General disorders) | 2
Peripheral swelling (General disorders) | 1
Pyrexia (General disorders) | 1
Thirst (General disorders) | 5
Hepatic function abnormal (Hepatobiliary disorders) | 3
Hypersensitivity (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 2
Bronchitis (Infections and infestations) | 3
Candida infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pharyngotonsillitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 6
Contusion (Injury, poisoning and procedural complications) | 2
Excoriation (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 3
Head injury (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood pressure decreased (Investigations) | 1
Blood urea increased (Investigations) | 1
Hepatic enzyme abnormal (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Weight decreased (Investigations) | 1
Weight increased (Investigations) | 19
White blood cell count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 9
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Increased appetite (Metabolism and nutrition disorders) | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Altered state of consciousness (Nervous system disorders) | 1
Amnesia (Nervous system disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 235
Dizziness postural (Nervous system disorders) | 7
Dysarthria (Nervous system disorders) | 1
Dyskinesia (Nervous system disorders) | 1
Dysstasia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 10
Hyperaesthesia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 2
Migraine (Nervous system disorders) | 1
Monoplegia (Nervous system disorders) | 1
Myoclonus (Nervous system disorders) | 1
Neuroleptic malignant syndrome (Nervous system disorders) | 1
Radicular pain (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 134
Transient ischaemic attack (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 3
Hallucination, auditory (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 7
Sleep disorder (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 4
Ureterolithiasis (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 2
Fixed eruption (Skin and subcutaneous tissue disorders) | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Skin erosion (Skin and subcutaneous tissue disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 3
Hot flush (Vascular disorders) | 4
Hypertension (Vascular disorders) | 4
Phlebitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2013-04-08): https://cdn.clinicaltrials.gov/large-docs/93/NCT01256593/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT01256593/SAP_001.pdf